CLINICAL TRIAL: NCT02021071
Title: Evaluation of Adding Virtual Path Planning to the Philips FD20 XperGuide to Reduce Radiation Dose During Image-guided Needle Interventional Procedures.
Brief Title: Virtual Path Planning for Image-guided Needle Interventions
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: XCY612-130031
Record Dates: First submitted 2013-11-27; First posted 2013-12-27 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Diseases; Bone Diseases; Muscular Diseases; Spinal Diseases; Vascular Diseases
MeSH Terms: conditions — Gastrointestinal Diseases; Bone Diseases; Muscular Diseases; Spinal Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- XperGuide: Image-guided needle procedures with XperGuide performed prior to this study within institution (retrospective data).
  Interventions: Radiation: XperGuide
- XperGuide with virtual path planning: Image-guided needle procedures with XperGuide with virtual path planning
  Interventions: Radiation: XperGuide with virtual path planning

INTERVENTIONS:
Radiation: XperGuide — Live 3D image needle guidance which overlays live fluoroscopy and 3D soft tissue imaging data from previous acquired CT, MR or XperCT.
  Groups: XperGuide
Radiation: XperGuide with virtual path planning — Instrument guidance allowing certain tasks that would normally occur using continuous X-ray guidance to be performed with reduced dose for patient and staff.
  Groups: XperGuide with virtual path planning

SUMMARY:
Philips Healthcare has added a virtual path planner to the current commercially available XperGuide software platform and that has the potential to significantly reduce dose during image-guided needle interventions.

DETAILED DESCRIPTION:
The investigational device is used for image guidance by virtually planned path and X-ray data.

ELIGIBILITY:
Inclusion Criteria:

* Patients at any age who are referred for a clinically indicated XperGuide interventional procedure.
* The informed consent has been signed by the participant, parent or legal guardian as appropriate.

Exclusion Criteria:

-Pregnant patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages. Patient weight is limited to the specification of the patient table.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Racadio, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of patients occurred between December 3rd 2013 and June 9th 2014.
Period: Overall Study
Arm/Group | XperGuide | XperGuide With Virtual Path Planning
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XperGuide | XperGuide With Virtual Path Planning | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Number; unit: participants]
  Newborn (birth - 1st month) | 0 | 0 | 0
  Infant (1st month - 2 years) | 0 | 0 | 0
  Child (2 - 12 years) | 2 | 2 | 4
  Adolescent (12-21 years) | 6 | 6 | 12
  Adult (> 21 years) | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (SUS) Score as a Measure of Qualitative Clinical Usefulness
Description: Evaluate the workflow, usability, and clinical impact of device by assessing clinical outcome and success of the procedures.
  The SUS is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability developed by Brooke, J. The user needs to provide agreement or disagreement for the 10 statements. After the appearing of the SUS in literature and once part of the ISO standard ISO 9241 Part 11 it has become an industry standard and has been used for over 25 years to measure usability.
  The minimum score is 0 and the maximum core is 100. Analysis of 500 studies with SUS showed that the average SUS score is a 68. A SUS score above a 68 would be considered above average and anything below 68 is below average
Time Frame: Patients will be followed starting from the procedure until hospital discharge or until 2 weeks after date of procedure at the latest
Population: SUS Score is only assessed for new technology (arm/group: XperGuide with virtual path planning)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | XperGuide With Virtual Path Planning
Number analyzed (Participants) | 12
Scores on a scale | 76 (16)

2. Secondary Outcome: Fluoroscopy Time
Description: Measure fluoroscopy time (minutes) needed during needle interventional procedure and compare the collected results with existing data from needle interventional procedures performed using XperGuide alone.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | XperGuide | XperGuide With Virtual Path Planning
Number analyzed (Participants) | 12 | 12
Minutes | 1.31 [0.51 to 8.48] | 0.45 [0.03 to 3.49]

ADVERSE EVENTS:
Time Frame: During procedure
Arm/Group | XperGuide | XperGuide With Virtual Path Planning
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No